CLINICAL TRIAL: NCT01911416
Title: A Biomarker Study to Identify Predictive Signatures of Response to LDE225 (Hedgehog Inhibitor) In Patients With Resectable Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI67198
Record Dates: First submitted 2013-07-11; First posted 2013-07-30 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental): All participants on study
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225

SUMMARY:
Pancreatic cancer is considered a rare form of cancer with about 277,000 new cases diagnosed in 2008 world-wide, which is about 2.5% of all forms of cancer. However, pancreatic cancer is more common in developed countries where the rate of this tumor is on the rise compared to other types of cancer.

LDE225 is a new medicine that blocks a cellular pathway (called Hedgehog pathway) that is thought to be changed in some patients with pancreatic cancer. LDE225 is a medicine which has not been approved by the FDA for the treatment of people with your medical condition. The medicine being tested in this study is currently not "on the market" (available to buy) in any country.

The purpose of this study is to see the effect LDE225 has on blood and tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically documented diagnosis of pancreatic ductal adenocarcinoma
* Patients with resectable pancreatic ductal adenocarcinoma or borderline resectable disease that after neoadjuvant treatment are considered appropriate candidates for resection
* ECOG or Performance Status of 0-2
* Patients with adequate bone marrow, liver and renal function, as specified below:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 80 x 109/L
  * Serum total bilirubin ≤ 1.5 x ULN(upper limit of normal)
  * AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present
  * Plasma creatine phosphokinase (CK) < 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50ml/min
* Written informed consent obtained prior to any study specific screening procedures

Exclusion Criteria:

* Patients who have had major surgery within 4 weeks of initiation of study medication.
* Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data.
* Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes.
* Patients who have previously been treated with systemic LDE225 or with other Hh pathway inhibitors.
* a) Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 2 weeks prior to starting LDE225 treatment. If it is essential that the patient stays on a statin to control hyperlididemia, only pravastatin may be used with extra caution. b) Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment. NB: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided whilst on LDE225 treatment.
* Patients who have taken part in an experimental drug study within 4 weeks of initiating treatment with LDE225.
* Patients who are receiving other anti-neoplastic therapy (e.g. chemotherapy, targeted therapy or radiotherapy) concurrently or within 2 weeks of starting treatment with LDE225.
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include:

  • Diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Reliable contraception should be maintained throughout the study and for 3 months after study drug discontinuation.
* Patients unwilling or unable to comply with the protocol.
* Patients who are not candidates to undergo laparoscopic examination and biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 36 months
  Correlation between plasma and tumour concentrations of LDE225

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garrido-Laguna, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States